CLINICAL TRIAL: NCT03692585
Title: Digitally Supporting Lifestyle Changes in Men With Prostate Cancer, Based on Characteristics and Needs - Part 1: Ethnographic Study of the Everyday Life of Men With Prostate Cancer, Focusing on Diet, Activities and Digital Behavior
Brief Title: Ethnographic Study of the Everyday Life of Men With Prostate Cancer, Focusing on Diet, Activities and Digital Behavior
Acronym: EMIL
Status: Completed | Type: Observational
Sponsor: Danish Cancer Society (Other)
Collaborators: University of Copenhagen (Other); TrygFonden, Denmark (Industry)
Responsible Party: Principal Investigator, Dorthe Furstrand, Ph.d. fellow, MD, Danish Cancer Society
Other Study IDs: DCS-53232017-1; Tryg-7-12-0736 (Other: Trygfonden)
Record Dates: First submitted 2018-09-29; First posted 2018-10-02 (Actual); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Prostate Cancer; Computer Literacy; Health Behavior
Keywords: Ethnography; Health Informatics; Healthy Lifestyle; Patient Involvement; eHealth Literacy
MeSH Terms: conditions — Prostatic Neoplasms; Health Behavior; Patient Participation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an ethnographic study to investigate the competences and preferences in everyday living of men with prostate cancer, using participant observation and semi-structured interviews.

The study will work as the need assessment part of the emil project, which aims to design, develop, implement and evaluate a digital service to support a healthy lifestyle among men with prostate cancer.

DETAILED DESCRIPTION:
Data was collected between June 2015 and April 2016. The data set included 4 parts; introducing interviews, participant observation, concluding interviews and questionnaires.

The introducing interview is conducted as a semi-structured interview with an interview guide. An informal approach is chosen to help along the report needed for the participant observation. The interview is recorded.

During participant observations, the participant is accompanied by the researcher, as he goes about his daily life. The researcher is participating in his activities to the extend it is possible, carrying out spontaneous informal interviews along the way taking cues from the situation, as is inherent to the participation of the researcher during participant observations. Field jottings are done discretely, during breaks in the observation or afterwards, on dictaphone or computer, in order to keep the relation informal, and not redirect the attention to the fact that they were being observed.

The concluding interview is performed as a natural ending of the collaboration between researcher and participant. It is performed as a semi-structured interview with an interview guide, and the central point is to confirm and elaborate on findings of the observation. The interview is recorded.

Pictures are taken of relevant artefacts or sceneries through all visits between participant and researcher, with the consent of the participants. Pictures are a part of the dataset on equal terms with observational notes and interview transcriptions.

In the questionnaire, baseline information such as educational level and self-rated health is gathered along with measurement of eHealth literacy (eHLQ) and health literacy (HLQ), both multidimensional validated psychometric instruments with seven and nine dimensions respectively, in order to relate the demography of this first study to the later studies of the emil project. The questionnaire is not used in the analysis of this study.

All data is collected before beginning familiarization and analysis of data.

Data analysis and interpretation The data set is analyzed using an inductive thematic analysis as described by Braun and Clarke (2006). All interviews and observations are conducted by the first author. Interviews, both introducing and concluding, are transcribed verbatim except for parts not included in the dataset, such as parts where the formal information about the study is given and written consent obtained or parts where practical arrangements are made.

All observational data are written together in one document from each visit. All pictures are included in the dataset. Familiarization with the data will be by listening and relistenning, reading and rereading through the dataset.

The thematic analysis will be performed by coding, processing and interpretation of data using the qualitative research software Nvivo11. Codes are re-read, discussed in the research group, re-coded and themed as outlined by the phases of Braun and Clarke, ending up with a thematic map.

ELIGIBILITY:
Inclusion Criteria:

* Men with a history of prostate cancer, self-reported

Exclusion Criteria:

* Participants will be excused from participation if they do not have sufficient written and spoken Danish language skills for participation in the activities involved in the studies. The researcher will assess whether the participants have sufficient cognitive functions to participate in the study. The researcher can also judge from an ethical perspective that the participant, for reasons not stated in the protocol, should be excused from participation in the study.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Danish Population
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2015-06; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Identification of factors that influence healthy lifestyle practices related to diet and physical activity for men with prostate cancer, in their everyday life | Data collection: 11 months
  Factors will be identified by using Thematic analysis (Braun and Clarke, 2006) of ethnographic data, including interview transcriptions, observational notes, pictures and artefacts from the participant observation. All themes are based on identified categories and coding of observations, and are confirmed by supporting quotes.
  The primary outcomes will be obtained in a way that it can inform the design process in the second study of the emil-project.

SECONDARY OUTCOMES:
Identification of digital capabilities and attitude of men with prostate cancer, in their everyday life | Data collection: 11 months
  Digital capabilities and attitude will be examined as a specific part of the Thematic analysis (Braun and Clarke, 2006) of ethnographic data, including interview transcriptions, observational notes, pictures and artefacts from the participant observation. All themes are based on identified categories and coding of observations, and are confirmed by supporting quotes.
eHealth literacy evaluation | Data collection: 11 months
  eHealth literacy evaluated by use of the eHealth Literacy questionnaire (eHLQ) and findings related to observed digital behavior.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Tjønneland, MD PhD DMSc, Study Director — Danish Cancer Society Research Center; Lars Kayser, MD PhD, Study Chair — University of Copenhagen, Dept. of Public Health

IPD SHARING:
Plan to Share IPD: Undecided
It is a priority to protect the privacy of participant according to research ethics guidelines and GDPR. Participant data will only be shared in anonymized form and only in the extend demanded by a journal.